CLINICAL TRIAL: NCT04776564
Title: Effectiveness and Satisfaction With the Gottman 7 Principles Couple Enhancement Courses in Norway
Brief Title: Effectiveness and Satisfaction With the Gottman Couple Enhancement Course
Status: Completed | Type: Observational
Sponsor: Rune Zahl-Olsen (Other Government)
Responsible Party: Sponsor-Investigator, Rune Zahl-Olsen, Senior Researcher, Sorlandet Hospital HF
Organization: Sorlandet Hospital HF (Other Government)
Other Study IDs: NSD-461755
Record Dates: First submitted 2021-02-19; First posted 2021-03-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Couples
Keywords: Gottman seven principles couple enhancement program; Couple enhancement program; Couple satisfaction; Marital relationship

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Intensive courses: Participants on courses delivered within four days
  Interventions: Other: Participation in the couple enhancement program
- Long courses: Participants on courses delivered over minimum four weeks
  Interventions: Other: Participation in the couple enhancement program
- Clinical: Participants attending G7P courses delivered within the specialist health care setting
  Interventions: Other: Participation in the couple enhancement program
- Internett: Participants attending G7P courses delivered as an online course
  Interventions: Other: Participation in the couple enhancement program
- Professional: Participants attending G7P courses wihere professional health care personell are delivering the teaching
  Interventions: Other: Participation in the couple enhancement program
- Non-professional: Participants attending G7P courses wihere no professional health care personell are delivering the teaching
  Interventions: Other: Participation in the couple enhancement program
- Control group: A sample of couples from the public that do not at the moment participate in couple therapy or any couple enhancement programs

INTERVENTIONS:
Other: Participation in the couple enhancement program — Participation in a 12 hour long couple enhancement program called Gottman seven principles (G7P)
  Groups: Clinical; Intensive courses; Internett; Long courses; Non-professional; Professional

SUMMARY:
This project will investigate the Gottman 7 principle couple course (G7P) in the Norwegian setting offered at different sites and for different groups of the population.

A control group of couples will serve as a baseline.

The study will bring knowledge about the participants experiences with the G7P and the effectiveness of the course on improving the couple relationship.

DETAILED DESCRIPTION:
This project will investigate the Gottman 7 principle couple course (G7P) in the Norwegian setting offered at different sites and for different groups of the population, including a sample of clients from the specialist health services. A control group of couples will serve as a baseline. The study will bring knowledge about the participants experiences with the G7P and the effectiveness of the course on improving the couple relationship.

The G7P couple enhancement program is translated to Norwegian and 200 trainers were licensed in 2017. Some of these trainers are professionals, such as psychologists and couple and family therapists and some are non-professionals. The courses are offered in communities all over the country and also for clients in specialized health care at Sorlandet hospital.

This project has a mixed-method design and will explore these research questions:

1. Do Gottman 7 principles courses lead to better couple functioning from start to end of program and at 6 months follow up? And if so, for whom?
2. Do different populations benefit equally from the course?
3. Who join Gottman 7p courses?
4. Why do they join a Gottman 7p course?
5. Is there any difference in the experience of the course and the effectiveness of the course when a professional or a non-professional is the trainer?
6. How do the participants experience the course and the usefulness of it?

Method:

To answer our research questions we want to obtain data through questionnaires and interviews, thus a mixed-method study. The project is a cohort study with three measurement points for the quantitative part and two for the qualitative part of the study. A control group of couples will serve as a baseline.

Quantitative sub-study:

Participants at G7P courses in Norway will be asked to participate in the quantitative part of the study. The participants are asked to answer some questions at the start and at the end of the course (t1, and t2) and six months after the course (t3).

Additional, a control group will participate in the study. They will be asked to participate through a) the Solide Samliv webpage and b) the Solide Samliv facebook page. c) advertizement on social media. The control group will answer to questions equal to t1 and t3.

Analyzes will be performed in SPSS, Jasp and R and both frequentist and Bayesian approaches will be used.

Qualitative sub-study:

This sub-study amnswers to research question 6: How do the participants experience the Gottman 7 principles course and the usefulness of it? Recruitment will take place through the G7P courses. The sample is recruited from those who signed the consent to participate in the study at the start of each course. The selection of participants will be based on variation in terms of informants' background (e.g. gender, age, length of the relationship, urban/rural), to illuminate the breadth of bereaved individuals' experiences. We are aiming at 18 participants. The sample shall consist of 6 men, 6 women, and 6 couples. Qualitative interviews will be conducted at two times: approximately at the end of the course and six months after the end of the course.

Data and method of collection: In-depth interviews will take place in part individually and in part as couples in a place chosen by the participants. The interview will be recorded by the researcher and then transcribed by external assistance.

Analysis: Thematic analysis of qualitative data (Clarke & Braun, 2014).

ELIGIBILITY:
Inclusion Criteria:

* Participating in a G7P course

Exclusion Criteria:

* None, except for if they do not sign the consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample and adult clients in specialist health care services wanting to strengthen their couple relationship
Sampling Method: Non-Probability Sample
Enrollment: 732 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Change in Dyadic Adjustment from baseline to the end of the course | Before the course start (Baseline, t0) and within one week after the last day of the course (t1)
  The Revised Dyadic Adjustment Scale (RDAS - (Busby et al., 1995) is a self-report questionnaire with 14 items.
  The three sub-scales (Consensus, Satisfaction and Cohesion) and the Total-scale will be used as outcome measures
  The min and max values are:
  Consensus [0-30] Satisfaction [0-20] Cohesion [0-19] Total scale [0-69]
  Higher values indicate better adjustment and clinical cut-off has been identified at 47.31 for the total scale, indicating a level of severity equal to what is found in clinical samples (persons seeking couple therapy).
Change in Dyadic Adjustment from the end of the course to 6 months after the course | Within one week after the last day of the course (t1) to six month after the course is finished (t2)
  The Revised Dyadic Adjustment Scale (RDAS - (Busby et al., 1995) is a self-report questionnaire with 14 items.
  The three sub-scales (Consensus, Satisfaction and Cohesion) and the total scale will be used as outcome measures.
  The min and max values are:
  Consensus [0-30] Satisfaction [0-20] Cohesion [0-19] Total scale [0-69]
  Higher values indicate better adjustment and clinical cut-off has been identified at 47.31 for the total scale, indicating a level of severity equal to what is found in clinical samples (persons seeking couple therapy).

SECONDARY OUTCOMES:
Change in couple satisfaction from baseline to the end of the course, with response shift. | Before the course start (t0) and within one week after the last day of the course (t1)
  Before the course start the participants assess their couple satisfaction on a single scale from 1 (very dissatisfied) to 5 (very satisfied). At the end of the course they are asked the same question.
  Additionally, at the end of the course, they are asked how they now, after participating in the course, would rate their couple satisfaction at the start (1-5). This provide us with a response shift perspective.
  Change will be assessed by comparing the change in the scores from start (t0) to end (t1), and by assessing the response shift (t0r).I.e. difference in perception from t0 and t0r and change in score from t0r to t1.
  Higher values are better, indicating a more satisfied relationship
Change in couple satisfaction from the end of the course to 6 months after the course | Within one week after the last day of the course (t1) to six month after the course is finished (t2)
  The participants assess their couple satisfaction on a single scale from 1 (very dissatisfied) to 5 (very satisfied).
  Change will be assessed by comparing the change in the scores from the end of the course (t1) to six months after the course (t2).
  Higher values are better, indicating a more satisfied relationship

CONTACTS AND LOCATIONS:
Overall Officials: Rune Zahl-Olsen, Principal Investigator — Senior researcher at Sørlandet Hospital HF
Locations (1):
- Sørlandet Hospital HF, Kristiansand, Agder, Norway

IPD SHARING:
Plan to Share IPD: Yes
After the data are analyzed the data and the code is planed to be shared with researchers of interest
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: By summer 2023 and until end of 2028 all this will be available, on request. However, some variables will be masked so that persons within the dataset cannot be identified using this data in combination of data elsewhere. This is information like the exact date and place of the course they attended.
Access Criteria: Serious researchers with plan for publishing or controll of the analysis will be given access.